CLINICAL TRIAL: NCT04345406
Title: Randomized Trial of ACEIs in Treatment of COVID-19
Brief Title: Angiotensin Converting Enzyme Inhibitors in Treatment of Covid 19
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, assistant professor of tropical medicine and infectious diseases, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACEIS COVID 19
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: COVID
MeSH Terms: interventions — Enalapril; Captopril; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEIs (Experimental): ACEIs with conventional treatment for COVID19
  Interventions: Drug: ACEIs; Drug: Conventional treatment
- Conventional treatment of COVID19 (Experimental): Conventional treatment of COVID19
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: ACEIs — Captopril or enalapril
  Other Names: Enalapril, Captopril
  Arms: ACEIs
Drug: Conventional treatment — alexoquine
  Other Names: chloroquine

SUMMARY:
ACEIs as treatment for COVID19

DETAILED DESCRIPTION:
ACEIs as suggested treatment for COVID19

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with covid 19

Exclusion Criteria:

* allergy or contraindications to the drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with virological cure | 6 months
  number of patients with virological cure

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, ass. prof., Principal Investigator — Tanta University Faculty of medicine
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No